CLINICAL TRIAL: NCT01425515
Title: Heart Healthy Lenoir: Improving Care for Patients With High Blood Pressure
Brief Title: Improving Care for Patients With High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jacquie Halladay, MD, MPH, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0395; P50HL105184 (NIH)
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension; Cardiovascular Disease Risk
Keywords: hypertension; genomics
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Complex quality improvement intervention — We are implementing a complex quality improvement intervention that includes changes in practice processes to enhance hypertension care, provision of home blood pressure monitors to patients, and telephone coaching around hypertension self-management.

SUMMARY:
The investigators are conducting a single group intervention study to improve blood pressure control and reduce racial and literacy related disparities among people with hypertension. The intervention includes providing patients with home blood pressure monitors, administering phone-coaching to participants, and improving hypertension care at the participating practices from which patients are enrolled. The investigators will follow the patients for 2 years to determine if blood pressure control improves. In addition, the project will explore genetic factors associated with cardiovascular disease risk and treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who meet the following inclusion criteria will be eligible for study participation:
* 18 years or older,
* Able and willing to give informed consent,
* A current patient of 1 of the 5 participating practices,
* Have a current diagnosis of hypertension by their primary care physician or have 3 documented blood pressures above 150/90,
* Their most recent systolic blood pressure was greater than or equal to 150 at their most recent clinic visit,
* Receive physician approval to participate in the study.
* Anyone enrolled in the High Blood Pressure study is eligible to participate in the genomics component of the project.

Exclusion Criteria:

* non-English speaking,
* current treatment of psychosis,
* diagnosed with advanced dementia as determined by the clinician,
* current substance abuse,
* lack of phone access,
* history of malignancy, other than non-melanoma skin cancer, that has not been in remission or cured surgically for > 5 years,
* estimated creatinine clearance less than 30 ml/min (because hypertension management becomes more complicated at this point),
* are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | 2 years
  We will measures blood pressure at enrollment and then every 6 months for 24 months.

SECONDARY OUTCOMES:
Blood lipids | 2 years
  We will measure blood lipids including total cholesterol and HDL over the course of the study to calculate overall cardiovascular risk.
General Cardiovascular Disease Risk | 2 years
  We will measure variables (blood pressure, cholesterol, aspirin use, smoking status, and diabetes status) to calculate general cardiovascular disease risk which includes (coronary death, myocardial infarction, coronary insufficiency, angina, ischemic stroke, hemorrhagic stroke, transient ischemic attack, peripheral artery disease, heart failure). (D'Agostino, 2008)
Genomic predictors of blood pressure change | 6-, 12-, 18, and 24-month follow-up
  A systems approach to developing genomic models integrating clinical and genomic data.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Halladay, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Kinston Enterprise Center - Study Office, Kinston, North Carolina, United States

REFERENCES:
- [Background] D'Agostino RB Sr, Vasan RS, Pencina MJ, Wolf PA, Cobain M, Massaro JM, Kannel WB. General cardiovascular risk profile for use in primary care: the Framingham Heart Study. Circulation. 2008 Feb 12;117(6):743-53. doi: 10.1161/CIRCULATIONAHA.107.699579. Epub 2008 Jan 22. PMID 18212285
- [Derived] Cummings DM, Adams A, Halladay J, Hinderliter A, Donahue KE, Cene CW, Li Q, Miller C, Garcia B, Tillman J, Little E, DeWalt D. Race-Specific Patterns of Treatment Intensification Among Hypertensive Patients Using Home Blood Pressure Monitoring: Analysis Using Defined Daily Doses in the Heart Healthy Lenoir Study. Ann Pharmacother. 2019 Apr;53(4):333-340. doi: 10.1177/1060028018806001. Epub 2018 Oct 3. PMID 30282468
- [Derived] Chatterjee A, Daftary G, Gatison L, Gillman MW. Lessons Learned From a Partnership to Evaluate a School Food Program. Prog Community Health Partnersh. 2016;10(4):577-584. doi: 10.1353/cpr.2016.0066. PMID 28569683
- [Derived] Cummings DM, Wu JR, Cene C, Halladay J, Donahue KE, Hinderliter A, Miller C, Garcia B, Penn D, Tillman J, DeWalt D. Perceived Social Standing, Medication Nonadherence, and Systolic Blood Pressure in the Rural South. J Rural Health. 2016 Spring;32(2):156-63. doi: 10.1111/jrh.12138. Epub 2015 Sep 3. PMID 26334761
- [Derived] Halladay JR, Donahue KE, Hinderliter AL, Cummings DM, Cene CW, Miller CL, Garcia BA, Tillman J, DeWalt D; Heart Healthy Lenoir Research Team. The Heart Healthy Lenoir project--an intervention to reduce disparities in hypertension control: study protocol. BMC Health Serv Res. 2013 Oct 25;13:441. doi: 10.1186/1472-6963-13-441. PMID 24156629
- See also: Summary information about the Heart Healthy Lenoir Project — http://hpdp.unc.edu/research/projects/heart-healthy-lenoir/